

16<sup>th</sup> October 2022

Mr. Wang Shaoshen Biostatistics and Research Methodology Unit School of Medical Sciences Universiti Sains Malaysia 16150 Kubang Kerian, Kelantan. Jawatankuasa Etika Penyelidikan Manusia USM (JEPeM)

Human Research Ethics Committee USM (HREC)

Universiti Sains Malaysia Kampus Kesihatan

16150 Kubang Kerian, Kelantan, Malaysia. Tel.: +609 - 767 3000/2354/2362

Fax. : + 609 - 767 2351 Email : jepem@usm.my

Laman Web : www.jepem.kk.usm.my

www.usm.mv

JEPeM Code: USM/JEPeM/22050298

Protocol Title: A Structural Equation Model and Effects of Music on Mental Energy, Mindfulness, Psychological Skills and Sports Performance among Young Basketball Players in Shandong Province, China.

Dear Mr.,

We wish to inform you that your study protocol has been reviewed and is hereby granted approval for implementation by the Jawatankuasa Etika Penyelidikan Manusia Universiti Sains Malaysia (JEPeM-USM). Your study has been assigned study protocol code USM/JEPeM/22050298, which should be used for all communications to JEPeM-USM in relation to this study. This ethical approval is valid from 16<sup>th</sup> October 2022 until 15<sup>th</sup> October 2023.

Study Site: Shandong Province, China.

The following researchers are also involved in this study:

- 1. Dr. Kueh Yee Cheng
- 2. Assoc. Prof. Dr. Garry Kuan Pei Ern
- 3. Assoc. Prof. Dr. Najib Majdi Yaacob

The following documents have been approved for use in the study.

1. Research Proposal

In addition to the abovementioned documents, the following technical documents were included in the review on which this approval was based:

- 1. Parental Information Sheet and Consent Form (English version)
- 2. Parental Information Sheet and Consent Form (Chinese version)
- 3. Feeling Scale (FS)
- 4. Athletic Mental Energy Scale (AMES)
- 5. The Brunel Mood Scale (BRUMS)
- 6. Felt Arousal Scale (FAS)
- 7. Athletic Identity Measurement Scale-Plus

The list of JEPeM-USM members present during the full board meeting reviewing your protocol is attached.

While the study is in progress, we request you to submit to us the following documents:

- Application for renewal of ethical approval 60 days before the expiration date of this approval through submission of JEPeM-USM FORM 3(B) 2019: Continuing Review Application Form.
- Any changes in the protocol, especially those that may adversely affect the safety of the participants during the conduct of the trial including changes in personnel, must be submitted or reported using JEPeM-USM FORM 3(A) 2019: Study Protocol Amendment Submission Form.



- 3. Revisions in the informed consent form using the JEPeM-USM FORM 3(A) 2019: Study Protocol Amendment Submission Form.
- 4. Reports of adverse events including from other study sites (national, international) using the JEPeM-USM FORM 3(G) 2019: Adverse Events Report.
- 5. Notice of early termination of the study and reasons for such using **JEPeM-USM FORM 3(E) 2019.**
- 6. Any event which may have ethical significance.
- 7. Any information which is needed by the JEPeM-USM to do ongoing review.
- 8. Notice of time of completion of the study using **JEPeM-USM FORM 3(C) 2019: Final Report Form.**

Please note that forms may be downloaded from the JEPeM-USM website: <a href="https://www.jepem.kk.usm.my">www.jepem.kk.usm.my</a>

JEPeM-USM is in compliance with the Declaration of Helsinki, International Conference on Harmonization (ICH) Guidelines, Good Clinical Practice (GCP) Standards, Council for International Organizations of Medical Sciences (CIOMS) Guidelines, World Health Organization (WHO) Standards and Operational Guidance for Ethics Review of Health-Related Research and Surveying and Evaluating Ethical Review Practices, EC/IRB Standard Operating Procedures (SOPs), and Local Regulations and Standards in Ethical Review.

Thank you.

"WAWASAN KEMAKMURAN BERSAMA 2030"

"BERKHIDMAT UNTUK NEGARA"

Sincerely,

DR. NOOR AMAN A. HAMID

Deputy Chairperson Jawatankuasa Etika Penyelidikan (Manusia), JEPeM Universiti Sains Malaysia



Date of meeting : 6<sup>th</sup> July 2022

Venue : Through WEBEX Application

Time : 9.00 a.m - 2.00 p.m

Meeting No : 550

Jawatankuasa Etika Penyelidikan Manusia USM (JEPeM)

Human Research Ethics Committee USM (HREC)

Universiti Sains Malaysia Kampus Kesihatan

16150 Kubang Kerian, Kelantan, Malaysia. Tel.: +609 - 767 3000/2354/2362

Fax. : + 609 - 767 2351 Email : jepem@usm.my

Laman Web : www.jepem.kk.usm.my

www.usm.my

Members of Committee of the Jawatankuasa Etika Penyelidikan (Manusia), JEPeM Universiti Sains Malaysia who reviewed the protocol/documents are as follows:

| | Member<br>(Title and Name) | Occupation<br>(Designation) | Male/<br>Female<br>(M/F) | Tick (✓) present<br>during review<br>process |
|---|---|---|---|---|
| <b>Deputy Chairperson:</b><br>Dr. Noor Aman A. Hamid | | Deputy Chairperson of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | M | √<br>(Deputy<br>Chairperson) |
| Advisor:<br>Professor Dr. Hans Amin Van Rostenberghe | | Advisor of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | М | √<br>(Advisor) |
| Advisor:<br>Assoc. Prof. Siti Hawa Ali | | Advisor of Jawatankuasa Etika<br>Penyelidikan (Manusia), JEPeM USM | F | √<br>(Advisor) |
| Secretary:<br>Mr. Mohd Bazlan Hafidz Mukrim | | Senior Science Officer | М | <b>✓</b> |
| Secretariat:<br>Miss Siti Fatihah Ariffin | | Research Officer | F | <b>√</b> |
| Memb | ers: | | | |
| 1. | Assoc. Prof. Dr. Garry Kuan Pei Ern | Lecturer, School of Health Sciences | М | ✓ |
| 2. | Prof. Dato' Dr. Jafri Malin Abdullah | Lecturer, School of Medical Sciences | М | <b>✓</b> |
| 3. | Dr. Khairil Amir Sayuti | Lecturer, School of Medical Sciences | М | <b>✓</b> |
| 4. | Prof. Dr. Mohtar Ibrahim | Lecturer, School of Medical Sciences | M | <b>✓</b> |
| 5. | Mrs. Normah Salleh | Community Representatives | F | <b>✓</b> |
| 6. | Prof. Dr. Oleksandr Krasilshchikov | Lecturer, School of Health Sciences | M | <b>✓</b> |
| 7. | Assoc. Prof. Dr. Saedah Ali | Lecturer, School of Medical Sciences | F | <b>✓</b> |
| 8. | Mrs. Zawiah Abu Bakar | Community Representatives | F | ✓ |
| 9. | Dr. Zuliani Mahmood | Lecturer, School of Dental Sciences | F | |

Jawatankuasa Etika Penyelidikan (Manusia), JEPeM-USM is in compliance with the Declaration of Helsinki, International Conference on Harmonization (ICH) Guidelines, Good Clinical Practice (GCP) Standards, Council for International Organizations of Medical Sciences (CIOMS) Guidelines, World Health Organization (WHO) Standards and Operational Guidance for Ethics Review of Health-Related Research and Surveying and Evaluating Ethical Review Practices, EC/IRB Standard Operating Procedures (SOPs), and Local Regulations and Standards in Ethical Review.



**DR. NOOR AMAN A. HAMID**Deputy Chairperson
Jawatankuasa Etika Penyelidikan (Manusia), JEPeM
Universiti Sains Malaysia